CLINICAL TRIAL: NCT05831878
Title: Disitamab Vedotin (RC48-ADC) in Patients With HER2-low Advanced Breast Cancer
Brief Title: RC48-ADC in HER2-low Advanced Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2023-054-B
Record Dates: First submitted 2023-04-16; First posted 2023-04-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — disitamab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC (Experimental): RC48-ADC as salvage treatment for HER2-low advanced breast cancer
  Interventions: Drug: Disitamab vedotin

INTERVENTIONS:
Drug: Disitamab vedotin — 2.0mg/kg, iv, day1, every 2 weeks
  Other Names: RC48-ADC

SUMMARY:
To evaluate the efficacy and safety of Disitamab vedotin (RC48-ADC) as salvage treatment in patients with HER2-low advanced breast cancer who have received up to one previous chemotherapy for recurrent or metastatic disease without previous use of antibody-drug conjugate.

DETAILED DESCRIPTION:
Subjects with HER2-low advanced breast cancer were treated with Disitamab vedotin as salvage treatment. ORR, PFS, OS and AE were assessed during the trial. HER2-low status is defined as IHC1+ or IHC2+ with negative FISH test.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years
* Expected survival ≥12 weeks
* ECOG 0-1
* Histologically confirmed invasive advanced or metastatic breast cancer that is incurable and unresectable
* At least one measurable lesion according to the RECIST 1.1
* No history of antibody-drug conjugate use
* Up to one previous chemotherapy for advanced disease
* Available hormone receptor status. Hormone receptor-positive subjects are allowed to receive no more than two previous endocrine therapy for advanced disease
* HER2-low tumors, defined as IHC1+ or IHC2+ with negative FISH test; or HER2-ultralow tumors, defined as incomplete and faint membrane staining in >0 but ≤10% of tumor cells
* Adequate organ function

Exclusion Criteria:

* History of thromboembolic events
* Uncontrolled systemic diseases, including diabetes, hypertension, interstitial lung disease, cirrhosis, etc.
* Active infections requiring systemic treatment
* Pregnant or lactating
* Presence of brain metastases and/or carcinomatous meningitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From the date of starting Disitamab Vedotin to the date of first documentation of progression or death (up to approximately 1 year)
  The percentage of subjects with complete remission (CR) or partial remission (PR) as the best response during the period from the beginning of the treatment to the progression of the disease or the completion of therapy (CR+PR)/Analysis of the total number of people.Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) was used to assess the objective tumor response.

SECONDARY OUTCOMES:
Adverse events | From the date of starting Disitamab Vedotin to the end of the treatment (up to approximately 1 year)
  Adverse events during Disitamab Vedotin regimen will be assessed according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, M.D., Principal Investigator — Renji Hospital,School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No